CLINICAL TRIAL: NCT06664814
Title: An Open-Label Phase 2 Study of N-Acetyl-D-Mannosamine (ManNAc) in Subjects With Primary Focal Segmental Glomerulosclerosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10002066; 002066-HG
Record Dates: First submitted 2024-10-26; First posted 2024-10-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-09

CONDITIONS: Focal Segmental Glomerulosclerosis
Keywords: FSGS; ManNAc; Sialic Acid; Proteinuria; Kidney Disease
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Proteinuria; Kidney Diseases | interventions — N-acetylmannosamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- open label, single arm (Experimental)
  Interventions: Drug: ManNAc

INTERVENTIONS:
Drug: ManNAc — 2 grams twice daily by mouth

SUMMARY:
Background:

Focal segmental glomerulosclerosis (FSGS) is a disease that causes scarring in parts of the kidneys that filter waste. This can lead to protein loss in the urine, which can worsen kidney function. The kidneys may fail over time, and dialysis or a kidney transplant may be needed. Other treatments for this disease do not always work and often have adverse effects. Better treatments for FSGS are needed.

Objective:

To test a study drug (ManNAc) in people with FSGS.

Eligibility:

People aged 18 years and older with FSGS.

Design:

Participants will have 5 to 6 clinic visits over 14 weeks. Two of the visits will require overnight stays for 2 or 3 nights.

ManNAc is a white powder that comes in a sachet. It is dissolved in water and taken twice a day by mouth. Participants will take their first dose at the clinic. They will learn how to store ManNAc and prepare each dose. They will record their doses in a diary. They will also write down any adverse effects or troubles they have using the drug at home.

During clinic visits, participants will have physical exams with blood and urine tests. They will complete questionnaires about their health, sleep habits, and fatigue symptoms.

During overnight visits, participants will also have 24-hour urine collection.

A study team member will call participants 1 week after the first dose to check on their health. Follow-up phone calls will then be every 2 weeks after each clinic visit.

Participants may meet with a dietitian to discuss nutrition while taking the ManNAc.

Participants may choose to have genetic tests.

DETAILED DESCRIPTION:
Study Description:

Phase 2, open-label, single-arm, single-center study of ManNAc 2,000 mg oral (PO) twice daily (BID) for 12 weeks in 15 subjects with primary focal segmental glomerulosclerosis (FSGS). The study will characterize the long-term safety, tolerability, pharmacokinetics, and efficacy of ManNAc for proteinuria reduction in subjects with primary FSGS. We hypothesize that ManNAc will be safe and well-tolerated and will reduce proteinuria in subjects with primary FSGS.

Objectives:

Primary Efficacy Objective:

Determine the efficacy of ManNAc therapy in reducing proteinuria in subjects with primary FSGS.

Primary Safety Objective:

Assess the long-term safety and tolerability of orally administered ManNAc to subjects with primary FSGS.

Secondary Objectives:

* Evaluate the long-term pharmacokinetic characteristics of ManNAc 2,000 mg PO BID administered to subjects with eGFR >=45ml/min/1.73msq.
* Evaluate the percent of subjects achieving partial or complete remission.

Exploratory Objectives:

* Evaluate the impact of ManNAc on symptom burden and functional status using patient-reported outcomes measures (PROMs).
* Evaluate the effect of ManNAc on clinical measures of renal function other than proteinuria.
* Evaluate the change in proteinuria as assessed by 24-hr urine collection.
* Assess variations in the clinical response to ManNAc therapy depending on whether glomerular hyposialylation is present or absent in pre-study renal biopsy samples.
* Assess variations in the clinical response to ManNAc therapy based on the presence of genetic variants in APOL1 in study subjects.

Endpoints:

Primary Endpoint:

Percentage reduction in proteinuria as assessed with urine protein/creatinine ratio (UPCR) from baseline through 12 weeks of ManNAc therapy.

Primary Safety Endpoint:

Demonstrate safety and tolerability by assessing the frequency of adverse events (AEs) in subjects as obtained from in-person assessments, clinical laboratory tests, vital signs, electronic diaries, and physical examinations.

Secondary Endpoints:

* To characterize plasma pharmacokinetics of ManNAc 2,000mg PO BID in subjects with eGFR >=45ml/min/1.73m^2.
* Proportion of FSGS patients meeting the FSGS Partial Remission of Proteinuria Endpoint (FPRE), defined as >40% UPCR reduction from baseline value and with an absolute value <1.5 g/g at the end of 12 weeks of therapy.
* Proportion of FSGS patients achieving complete remission (CR) defined as absolute value of UPCR <0.3 g/g at the end of 12 weeks of treatment.

Exploratory Endpoints:

* Change in PROMs as measured using the generic questionnaire Patient Reported Measurement Information System (PROMIS), from baseline to 12 weeks of ManNAc therapy.
* Change in eGFR slope of a linear regression line from baseline through 12 weeks.
* Proportion of FSGS patients with at least a 27% (geometric mean) reduction in urine albumin/creatinine ratio (UACR) from baseline values at end of 12 weeks of therapy.
* Reduction in 24-hr urine protein excretion from baseline after completion of ManNAc therapy at 12 weeks.
* Assess differences in endpoints based on the extent of glomerular hyposialylation in pre-study renal biopsy samples.
* Assess differences in endpoints based on presence of APOL1 genetic variants.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals must meet all the following inclusion criteria to be eligible to participate in this study:

* Prior kidney biopsy demonstrating FSGS obtained within 10 years prior to the screening visit.
* Age >=18 years weighing more than 50 kg.
* If the patient is on immunosuppressive therapy (e.g., prednisone, cyclosporine, tacrolimus or mycophenolate mofetil) he/she should be on these medications for at least 3 months prior to study evaluation and should be on a stable dose of the medication for at least 4 weeks before start of trial, with no plans to alter the regimen during 12 weeks of study period, except to stabilize levels and/or for any safety concerns.
* Subjects will be allowed to continue with standard of care (SOC) non-immunosuppressant antiproteinuric agents to include RAAS inhibitors, mineralocorticoid antagonists (MRA), sodium-glucose co-transporter-2 inhibitors (SGLT2i), non-dihydropyridine calcium channel blockers (NDHP-CCBs), and glucagon-like peptide-1 (GLP-1) receptor agonists, in addition to other SOC adjuvant therapies such as diuretics, if they are able to maintain a stable dose throughout the trial. Subjects and their primary nephrologists will be encouraged to optimize their SOC treatments as much as possible prior to trial commencement. Subjects must be on a stable dose for at least 4 weeks before start of trial. Subjects should attempt to keep stable doses of both immunosuppressants and anti-proteinuric drugs throughout trial duration, to avoid confounding effects. Patients not receiving any of these SOC agents either due to allergy or intolerance will still be eligible.
* Subjects must have a spot random urine PCR of >= 2g/g on each of 3 measurements collected on at least 2 separate days during screening period plus a 24-hr urine protein collection of >= 2g/day. The rationale for using this degree of proteinuria is that proteinuria beyond this threshold value significantly increases the risk of progressive decline of renal functions in the absence of effective therapies to mitigate this risk. Conversely, this threshold value could also allow for the selection of a cohort of patients who are most likely to benefit from ManNAc therapy.
* Subjects with an estimated glomerular filtration rate (eGFR) >=45 mL/min/1.73/m^2 using the race-free CKD-EPI 2021 equation based on creatinine and cystatin-C [Inker et al, 2021]. The rationale is that below this eGFR threshold, sialic acid, the key metabolite of ManNAc markedly accumulates and may potentially result in systemic toxicity. Prior pharmacokinetic studies have shown that renal elimination of sialic acid is primarily through glomerular filtration, and it is neither reabsorbed nor secreted in the renal tubules. Hence decline in eGFR below 45 mL/min/1.73m^2 directly correlates with rising blood sialic acid levels [Fuentes et al, 2020], in addition, these subjects may not benefit as much from ManNAc therapy as they have advanced disease pathology, which may be irreversible. Future studies with personalized precision ManNAc dosing may benefit the patient population with eGFR <45 mL/min/1.73m^2.
* Subjects of reproductive potential must be willing to use at least one effective form of birth control throughout the trial period, unless they have had a permanent birth control procedure/intervention including but not limited to hysterectomy, tubal ligation and/or vasectomy. These may include the following: barrier methods (such as condoms), oral or depot injection (for example, Norplant or Depo-Provera) contraception medication, and/or intrauterine devices.
* Evidence of a personally signed and dated informed consent indicating that the patient has been informed of all pertinent aspects of the study and their willingness to comply with all aspects of the study and their willingness to comply with all aspects of the study protocol, including treatment plan, laboratory tests, baseline and follow-up visits and procedures that include completion of daily diaries to record symptoms and medication intake.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Individuals who are unwilling or unable to provide informed consent.
* Individual presenting for initial therapy of uncontrolled nephrotic syndrome which we define as proteinuria as measured by spot urine protein:creatinine ratio >3g/g or 24-hour urine protein excretion of >3.5g/day with symptomatic peripheral edema or pulmonary edema, hypoalbuminemia (serum albumin <3.0g/dl), electrolyte disturbances (related or unrelated to medical therapy), and/or active thromboembolism (initiated on systemic anticoagulation in the last 3 months). The rationale for this criterion is that patient presenting for initial therapy for uncontrolled nephrotic syndrome may need to be initiated on various medications including immunosuppressives as well as non-immunosuppressive drugs which can significantly change the level of proteinuria. Additionally, fluid shifts due to diuretic use for treating edema can alter GFR which could confound the pharmacokinetics and pharmacodymanics of the investigational drug.
* Individuals who acutely require optimization of volume status with intravenous diuretics to control volume overload, as this may result in fluid shifts between the intravascular space and the remainder of extracellular fluid volume. This might alter drug pharmacokinetics and pharmacodynamics as mentioned above in # 2.
* Individuals with a psychiatric illness or neurological disease that in the judgement of the investigators would interfere with the ability to adhere with the requirements of this protocol. This includes, but is not limited to, uncontrolled/untreated psychotic depression, bipolar disorder, schizophrenia, substance abuse or dependence, antisocial personality disorder, panic disorder, or behavioral problems, which might interfere with effective communication.
* Vulnerable individuals, including those with impaired cognitive function or are incarcerated.
* Individuals whose renal biopsy shows evidence of an additional pathology along with FSGS.
* Renal biopsy showing interstitial fibrosis and tubular atrophy (IFTA) >50% per biopsy report.
* Individuals with uncontrolled hypertension with blood pressures consistently >140/90 mmHg on 3 or more community clinic blood pressure measurements.
* Individuals with clinical evidence of any type of active infection including but not limited to HIV, Hepatitis B and/or Hepatitis C or patients who are positive on screening test for HIV including antibody or viral load, HBV surface antigen and/or HCV antibody. If a patient is positive for HCV antibody, then an HCV viral load will be measured to identify subjects with active infection. Additional tests may include those to screen for active CMV, Infectious Mononucleosis (Epstein-Barr Virus), parvovirus B19 and/or COVID-19 infection as per investigator judgement.
* Individuals with evidence and/or documented history of progressive deterioration of liver functions, including the production of clotting factors, removal of toxic metabolic products, bile excretion for at least 6 months, routine hepatic laboratory indices including but not limited to (AST, ALT, or GGT) greater than 3 times the upper limit of normal, and/or individuals with a documented history and/or diagnosis of chronic liver disease.
* Individuals with hypertriglyceridemia >500 mg/dL.
* Individuals with a documented history of malignancy (identified in last 5 years or on active therapy at time of screening).
* Individuals with a documented history of Type I or Type II Diabetes Mellitus
* Individuals with documented history of hematological conditions commonly associated with FSGS such as sickle cell disease and myeloproliferative disorders.
* Individuals with a documented history of cardiac conditions commonly associated with FSGS such as congenital cyanotic heart disease. Individuals with a documented history of connective tissue disorders commonly associated with FSGS such as SLE and multiple sclerosis.
* Individuals taking medications (either currently or within the last 6 months) associated with FSGS such as interferons, lithium, androgenic steroids, sirolimus, heroin, anthracyclines and bisphosphonates.
* Individuals who are pregnant, will be breastfeeding or refuse birth control anytime during the study.
* Individuals who have received treatment with another investigational drug, investigational device, or approved therapy for investigational use less than 60 days prior to planned ManNAc dosing.
* Individuals with hypersensitivity to ManNAc.
* Individuals who have been treated with ManNAc, sialic acid, IVIG, and/or other supplements containing sialic acid (e.g., sialyllactose) less than 60 days prior to planned ManNAc dosing.
* Individuals who received a renal or any other solid organ and/or bone marrow/stem cell transplantation.
* Individuals who in the judgment of the investigator, have a condition that places the subject at increased risk for AEs or has any other illness or clinical condition that might confound the results of the study or pose an additional risk in administering study drug to the subject.
* Patients who need systemic immunosuppressive or glucocorticoid therapy for non-renal indication at any time throughout the trial.
* Any patient receiving rituximab, cyclosphosphamide and/or plasmapheresis within 6 months of screening.
* A documented history of active alcohol and/or substance abuse within the past 2 years.
* Any patient with collapsing FSGS variant on renal biopsy.
* Individuals with clinical history suggesting a post-adaptive FSGS such as those with neonatal history of low birth weight, congenital anomaly of the kidney or urinary tract (CAKUT) based on renal ultrasound findings or history of nephrectomy, vesicoureteral reflux or obesity as defined by Body Mass Index (BMI) > 40kg/m^2.

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Determine the efficacy of ManNAc therapy in reducing proteinuria in subjects with primary FSGS. | 12-weeks.
Assess the long-term safety and tolerability of orally administered ManNAc to subjects with primary FSGS. | 12-weeks.

SECONDARY OUTCOMES:
Evaluate the percent of subjects achieving partial or complete remission. | 12-weeks.
Evaluate the long-term pharmacokinetic characteristics of ManNAc. | 12-weeks.

CONTACTS AND LOCATIONS:
Overall Officials: William A Gahl, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
pending

REFERENCES:
- [Background] Galeano B, Klootwijk R, Manoli I, Sun M, Ciccone C, Darvish D, Starost MF, Zerfas PM, Hoffmann VJ, Hoogstraten-Miller S, Krasnewich DM, Gahl WA, Huizing M. Mutation in the key enzyme of sialic acid biosynthesis causes severe glomerular proteinuria and is rescued by N-acetylmannosamine. J Clin Invest. 2007 Jun;117(6):1585-94. doi: 10.1172/JCI30954. PMID 17549255
- [Background] Gelberg H, Healy L, Whiteley H, Miller LA, Vimr E. In vivo enzymatic removal of alpha 2-->6-linked sialic acid from the glomerular filtration barrier results in podocyte charge alteration and glomerular injury. Lab Invest. 1996 May;74(5):907-20. PMID 8642786
- [Background] Huizing M, Yardeni T, Fuentes F, Malicdan MCV, Leoyklang P, Volkov A, Dekel B, Brede E, Blake J, Powell A, Chatrathi H, Anikster Y, Carrillo N, Gahl WA, Kopp JB. Rationale and Design for a Phase 1 Study of N-Acetylmannosamine for Primary Glomerular Diseases. Kidney Int Rep. 2019 Jun 25;4(10):1454-1462. doi: 10.1016/j.ekir.2019.06.012. eCollection 2019 Oct. PMID 31701055
- [Background] Ito M, Sugihara K, Asaka T, Toyama T, Yoshihara T, Furuichi K, Wada T, Asano M. Glycoprotein hyposialylation gives rise to a nephrotic-like syndrome that is prevented by sialic acid administration in GNE V572L point-mutant mice. PLoS One. 2012;7(1):e29873. doi: 10.1371/journal.pone.0029873. Epub 2012 Jan 13. PMID 22253810
- [Background] Kakani S, Yardeni T, Poling J, Ciccone C, Niethamer T, Klootwijk ED, Manoli I, Darvish D, Hoogstraten-Miller S, Zerfas P, Tian E, Ten Hagen KG, Kopp JB, Gahl WA, Huizing M. The Gne M712T mouse as a model for human glomerulopathy. Am J Pathol. 2012 Apr;180(4):1431-40. doi: 10.1016/j.ajpath.2011.12.023. Epub 2012 Feb 7. PMID 22322304
- [Background] Niethamer TK, Yardeni T, Leoyklang P, Ciccone C, Astiz-Martinez A, Jacobs K, Dorward HM, Zerfas PM, Gahl WA, Huizing M. Oral monosaccharide therapies to reverse renal and muscle hyposialylation in a mouse model of GNE myopathy. Mol Genet Metab. 2012 Dec;107(4):748-55. doi: 10.1016/j.ymgme.2012.10.011. Epub 2012 Oct 18. PMID 23122659
- [Background] Pawluczyk IZ, Najafabadi MG, Brown JR, Bevington A, Topham PS. Sialic acid supplementation ameliorates puromycin aminonucleoside nephrosis in rats. Lab Invest. 2015 Sep;95(9):1019-28. doi: 10.1038/labinvest.2015.78. Epub 2015 Jun 29. PMID 26121320
- [Background] Troost JP, Trachtman H, Nachman PH, Kretzler M, Spino C, Komers R, Tuller S, Perumal K, Massengill SF, Kamil ES, Oh G, Selewski DT, Gipson P, Gipson DS. An Outcomes-Based Definition of Proteinuria Remission in Focal Segmental Glomerulosclerosis. Clin J Am Soc Nephrol. 2018 Mar 7;13(3):414-421. doi: 10.2215/CJN.04780517. Epub 2017 Nov 22. PMID 29167190
- [Background] Troost JP, Waldo A, Carlozzi NE, Murphy S, Modersitzki F, Trachtman H, Nachman PH, Reidy KJ, Selewski DT, Herreshoff EG, Srivastava T, Gibson KL, Derebail VK, Lin JJ, Hingorani S, Fornoni A, Fervenza FC, Sambandam K, Athavale AM, Kopp JB, Reich HN, Adler SG, Greenbaum LA, Dell KM, Appel G, Wang CS, Sedor J, Kaskel FJ, Lafayette RA, Atkinson MA, Lieske JC, Sethna CB, Kretzler M, Hladunewich MA, Lemley KV, Brown E, Meyers KE, Gadegbeku CA, Holzman LB, Jefferson JA, Tuttle KR, Singer P, Hogan MC, Cattran DC, Barisoni L, Gipson DS; Nephrotic Syndrome Study Network. The longitudinal relationship between patient-reported outcomes and clinical characteristics among patients with focal segmental glomerulosclerosis in the Nephrotic Syndrome Study Network. Clin Kidney J. 2019 Aug 5;13(4):597-606. doi: 10.1093/ckj/sfz092. eCollection 2020 Aug. PMID 32905199
- [Background] van der Willik EM, van Breda F, van Jaarsveld BC, van de Putte M, Jetten IW, Dekker FW, Meuleman Y, van Ittersum FJ, Terwee CB. Validity and reliability of the Patient-Reported Outcomes Measurement Information System (PROMIS(R)) using computerized adaptive testing in patients with advanced chronic kidney disease. Nephrol Dial Transplant. 2023 May 4;38(5):1158-1169. doi: 10.1093/ndt/gfac231. PMID 35913734
- [Background] Weinhold B, Sellmeier M, Schaper W, Blume L, Philippens B, Kats E, Bernard U, Galuska SP, Geyer H, Geyer R, Worthmann K, Schiffer M, Groos S, Gerardy-Schahn R, Munster-Kuhnel AK. Deficits in sialylation impair podocyte maturation. J Am Soc Nephrol. 2012 Aug;23(8):1319-28. doi: 10.1681/ASN.2011090947. Epub 2012 Jun 28. PMID 22745475
- [Derived] Huizing M, Ganguli A, Bolanos J, Leoyklang P, Wilkins KJ, Zeng Y, Figg WD, Rossignol F, Malicdan MCV, Kopp JB, Gahl WA; NIH-ManNAc Study Team. Phase 1 Study of Oral N-Acetylmannosamine in Primary Podocytopathies. Kidney Int Rep. 2025 Dec 31;11(3):103758. doi: 10.1016/j.ekir.2025.103758. eCollection 2026 Mar. PMID 41630898
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002066-HG.html